CLINICAL TRIAL: NCT04763694
Title: Dynamic Change in Accommodation After Wearing Multifocal Soft Contact Lenses for Myopia Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York College of Optometry (Other)
Responsible Party: Principal Investigator, Xiaoying Zhu, Assistant Clinical Professor, State University of New York College of Optometry
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRBNET ID 1325316
Record Dates: First submitted 2021-02-11; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Myopia; Accommodation
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment arm (Experimental): Subjects wore multifocal soft contact lenses for 12 months.
  Interventions: Device: Multifocal soft contact lenses

INTERVENTIONS:
Device: Multifocal soft contact lenses — Myopic subjects wore multifocal soft contact lenses for 12 months

SUMMARY:
The purpose of this study is to report the changes in accommodation, aberrations, and myopia in patients wearing multifocal soft contact lens for various durations.

The study objectives are to:

1. Determine the effects of wearing multifocal soft contact lens on accommodation and aberrations over a 12-month period.
2. Determine the effect of wearing multifocal soft contact lens on myopia over a 12-month period.

ELIGIBILITY:
Inclusion Criteria:

* Age: 8-17 years
* Refractive error: Sphere ≤ -10.00D, Cylinder ≤ 1.00D
* Monocular BCVA 20/25 or better
* No previous CL experience required

Exclusion Criteria:

* History of ocular pathology, binocular vision anomalies, refractive surgery, previous myopia control therapy, pharmaceutical agent known to affect accommodation.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-12-05 (Actual); Study Completion 2020-12-05 (Actual)

PRIMARY OUTCOMES:
Axial length | 12 months
  Change in axial length over the duration of the study
Refractive error | 12 months
  Change in refractive error over the duration of the study
Accommodation | 12 months
  Accommodation at various distances during the study

SECONDARY OUTCOMES:
Phoria | 12 months
  The amount of horizontal phoria (in prism diopter) at near while the subjects wore multifocal soft contact lenses, measured using Modified Thorington

CONTACTS AND LOCATIONS:
Overall Officials: Stewart Bloomfield, PhD, Study Director — State University of New York College of Optometry
Locations (1):
- State University of New York, New York, New York, United States